CLINICAL TRIAL: NCT05907382
Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of JMKX003002 in Single and Multiple Ascending Dose Randomized，Doubled-blind Phase 1 Study in Healthy Subjects
Brief Title: Safety, Tolerability of JMKX003002 in Phase 1 Study in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: JY-JM3002-101
Record Dates: First submitted 2023-05-23; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-05

CONDITIONS: Safety and Tolerability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- JMKX003002 SAD experimental group (Experimental): Participants will be randomized into 5 cohorts to receive single oral dose of JMKX003002 on Day 1. The doses in each cohort will be escalated based on the safety and pharmacokinetics (PK) / Pharmacodynamics (PD) data of the previous cohort.
  Interventions: Drug: JMKX003002 will be administered orally
- JMKX003002 MAD experimental group (Experimental): Participants will be randomized into 2 cohorts to receive orally twice -daily of JMKX003002 for 7 consecutive days. The second cohort will be escalated based on the safety and pharmacokinetics (PK)/ Pharmacodynamics (PD) data of the previous cohort.
  Interventions: Drug: JMKX003002 will be administered orally
- JMKX003002 FE experimental group (Experimental): Participants will receive 3 Sequence regimens, with a washout period between treatments.
  Interventions: Drug: JMKX003002 will be administered orally
- Placebo in Cohorts 1 to 5 (Placebo Comparator): Participants in Cohorts 1 to 5 will receive single oral dose of matching placebo on Day 1.
  Interventions: Drug: Placebo in Cohorts 1 to 5
- Placebo in 2 Cohorts (Placebo Comparator): Participants in 2 Cohorts will receive orally twice -daily of matching placebo for 7 consecutive days.
  Interventions: Drug: Placebo in 2 Cohorts

INTERVENTIONS:
Drug: JMKX003002 will be administered orally — oral once
  Other Names: JMKX003002
  Arms: JMKX003002 SAD experimental group
Drug: JMKX003002 will be administered orally — oral once
  Other Names: JMKX003002
  Arms: JMKX003002 MAD experimental group
Drug: JMKX003002 will be administered orally — oral once
  Other Names: JMKX003002
  Arms: JMKX003002 FE experimental group
Drug: Placebo in Cohorts 1 to 5 — oral once
  Other Names: Matching placebo will be administered orally
  Arms: Placebo in Cohorts 1 to 5
Drug: Placebo in 2 Cohorts — oral once
  Other Names: Matching placebo will be administered orally
  Arms: Placebo in 2 Cohorts

SUMMARY:
Safety, tolerability, pharmacokinetics, and pharmacodynamics of JMKX003002 in single and multiple ascending dose randomized，doubled-blind phase 1 study in healthy subjects

DETAILED DESCRIPTION:
Pharmacokinetic (PK) parameters, Pharmacodynamics

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18-45 years (inclusive);-
2. With normal or abnormal but clinically insignificant comprehensive physical examination (vital signs, physical examination), laboratory tests (hematology, blood biochemistry, urinalysis, coagulation function test) and, 12-lead ECG;
3. Subjects who understand study procedures and methods, voluntarily participate in this trial, follow study-related instructions, and sign a written informed consent form.

Exclusion Criteria:

1. Clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematologic, metabolic, endocrine, neurologic, psychiatric disease, or any condition that may interfere with the subject successfully completing the trial
2. Subjects with history of or current malignancy;
3. Participant who the researchers believe that there are volunteers who are not suitable for

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Number of the Adverse Events that are related to the single dose treatment | from baseline to Day 11
  single dose safety
Number of the Adverse Events that are related to the multiple dose treatment from baseline to Day 18 | from baseline to Day 18
  multiple dose safety

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital Fudan University, Shanghai, Shanghai Municipality, China